CLINICAL TRIAL: NCT01725685
Title: A Randomized, Double Blind, Single-dose, Three-period, Crossover Study to Investigate Pharmacokinetic, Safety and Tolerability of Fluticasone Furoate With Umeclidinium When Administered in Combination and as Monotherapies in Adult Healthy Volunteer Subjects
Brief Title: To Investigate the Pharmacokinetics and Safety of Fluticasone Furoate (FF)/ Umeclidinium (UMEC) Combination Compared With FF and UMEC Monotherapies in Adult Healthy Volunteers Using a Dry Powder Inhaler (DPI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 116524
Record Dates: First submitted 2012-11-01; First posted 2012-11-14 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: healthy volunteers; Umeclidinium; tolerability; Safety; Fluticasone Furoate; Pharmacokinetics
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A - FF 400 microgram (mcg) (Experimental): Subjects will be randomized to single dose of FF 400 mcg in either of the three treatment period, which is separated by a wash-out period of 7 to 10 days.
  Interventions: Drug: FF 400 mcg
- Treatment B - UMEC 500 mcg (Experimental): Subjects will be randomized to single dose of UMEC 125 mcg in either of the three treatment period, which is separated by a wash-out period of 7 to 10 days.
  Interventions: Drug: UMEC 500 mcg
- Treatment C - FF/UMEC 400/500 mcg (Experimental): Subjects will be randomized to single dose of FF/UMEC 100/125 mcg in either of the three treatment period, which is separated by a wash-out period of 7 to 10 days.
  Interventions: Drug: FF/UMEC 400/500 mcg

INTERVENTIONS:
Drug: FF 400 mcg — FF will be available as 100 mcg strength administered as 4 inhalations from a DPI
  Arms: Treatment A - FF 400 microgram (mcg)
Drug: UMEC 500 mcg — UMEC will be available as 125 mcg strength administered as 4 inhalations from a DPI
  Arms: Treatment B - UMEC 500 mcg
Drug: FF/UMEC 400/500 mcg — FF/UMEC will be available as 100/125 mcg strength administered as 4 inhalations from a DPI
  Arms: Treatment C - FF/UMEC 400/500 mcg

SUMMARY:
This will be a randomized, double-blind, single-dose, three-period balanced crossover study in adult healthy subjects. Each of the 18 subjects will be randomized to receive a treatment sequence consisting of each of the three treatments (FF 400 microgram (mcg), UMEC 500 mcg and FF 400 mcg/UMEC 500 mcg), in three consecutive periods, with a wash-out period of 7 to 10 days between the periods.

The study will include a Screening period (28 days prior to first dose), Treatment period (3 single dose periods separated by two 7 to 10 days washout periods) and Follow-up period (7 to 14 days post last dose).

The pharmacokinetic (PK) and safety assessments will be performed during the study at fixed timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GlaxoSmithKline (GSK) Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Child-bearing potential and is abstinent or agrees to use the contraception methods listed in Protocol for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow up visit (i.e. until after the follow up visit is complete; Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 million international units (MlU)/milliliter (ml) and estradiol <40 picograms (pg)/ml (<147 pmol/L) is confirmatory] Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use the contraception methods listed in Protocol if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status prior to study enrollment. For most forms of HRT, at least 2 to 4 weeks should elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
* Women who are confirmed postmenopausal or permanently sterilized (e.g. tubal occlusion, tubal ligation, hysterectomy, bilateral salpingectomy).
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Protocol. This criterion must be followed from the time of the first dose of study medication until the follow up visit.
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5xupper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Average QT duration corrected for heart rate by Fridericia's formula (QTcF) < 450 miliseconds (msec).
* Body mass index (BMI) within the range 19 to 33 kilogram (kg)/meter square (m2) (inclusive).
* Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of ≤10 pack years.[number of pack years = (number of cigarettes per day /20) x number of years smoked]

Exclusion Criteria

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* A positive pre-study drug/alcohol screen.
* A positive test for human Immunodeficiency virus (HIV) antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 mililitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of respiratory disease (i.e. history of asthmatic symptoms) in the last 10 years.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Unable to refrain from consumption of red wine, seville oranges, grapefruit or grapefruit juice and pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* Known or suspected sensitivity to the constituents of the DPI or a history of severe milk protein allergy.
* A supine mean heart rate outside the range 40 to 90 beats per minute (bpm) at screening.
* Diseases preventing use of anticholinergics: Diagnosis of narrow-angle glaucoma, or bladder neck obstruction that in the opinion of the study investigator or GSK medical monitor would pose a safety risk with use of an inhaled anticholinergic.
* Other concurrent diseases/abnormalities: A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the patient at risk through study participation if the condition/disease exacerbated during the study. The investigator is encouraged to contact the study medical monitor if further clarification is required.
* Affiliation with the investigators site

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2013-01-02 (Actual); Study Completion 2013-01-02 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) in plasma for FF and UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 5 minutes [mins], 15 mins, 30 mins, 45 mins, 1 hour (h), 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The PK parameter Cmax will be calculated for FF/UMEC in combination and as monotherapies
Area under the concentration-time curve (AUC(0-t)), where t is time of last measurable concentration in plasma for FF and UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The PK parameter AUC(0-t) will be calculated for will be calculated for FF/UMEC in combination and as monotherapies
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time [AUC(0-inf)] in plasma for FF and UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The PK parameter AUC(0-inf) will be calculated for will be calculated for FF/UMEC in combination and as monotherapies
Time of maximum observed concentration (tmax) in plasma for FF and UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Time of last measurable concentration (tlast) in plasma for FF and UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Plasma elimination half life (t½) in plasma for FF and UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Elimination rate constant (Lambda z) in plasma for FF and UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Apparent clearance (CL/F) in plasma for FF and UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Apparent volume of distribution (V/F) in plasma for FF and UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The FF and UMEC PK parameter in plasma will be calculated to compare the PK of FF/UMEC in combination with FF and UMEC monotherapies
Cumulative amount excreted drug in urine (Ae) for UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 0-6 h, 0-8 h, 0-12 h, 0-16 h) and Day 2(0-24 h)
  The UMEC PK parameter in urine will be calculated to compare the PK of UMEC when co-administered with FF; with UMEC as a monotherapy
Percent of dose excreted (% Fe) in urine for UMEC | Period 1, 2 and 3: Day 1 (pre-dose, 0-6 h, 0-8 h, 0-12 h, 0-16 h) and Day 2 (0-24 h)
  The UMEC PK parameter in urine will be calculated to compare the PK of UMEC when co-administered with FF; with UMEC as a monotherapy
Urine half life (urine t½) for UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 0-6 h, 0-8 h, 0-12 h, 0-16 h) and Day 2 (0-24 h)
  The UMEC PK parameter in urine will be calculated to compare the PK of UMEC when co-administered with FF; with UMEC as a monotherapy
Renal clearance (CLr) in urine for UMEC, if data permits | Period 1, 2 and 3: Day 1 (pre-dose, 0-6 h, 6-8 h, 8-12 h, 12-16 h) and Day 2(16-24 h)
  The UMEC PK parameter in urine will be calculated to compare the PK of UMEC when co-administered with FF; with UMEC as a monotherapy
Area under the concentration-time curve from time zero (pre-dose) to the time at which AUC is calculable for all subjects (AUC(0-t')), where t' is the time at which AUC is calculable for all the subjects | Period 1, 2 and 3: Day 1 (pre-dose, 5 mins, 15 mins, 30 mins, 45 mins, 1 h, 1.5 h, 2 h, 3 h, 4 h, 6 h, 8 h, 12 h, and 16 h) and Day 2 (24 h)
  The PK parameter AUC(0-t') will be calculated for will be calculated for FF/UMEC in combination and as monotherapies

SECONDARY OUTCOMES:
Clinical Safety data assessed as number of adverse events (AE) in each treatment group | Period 1 Day 1 dose to Follow up visit
  Safety and tolerability will be assessed by recording of AEs for subjects receiving FF/UMEC in combination compared with FF and UMEC monotherapies.
Clinical laboratory measurements for each treatment group | Period 1, 2 and 3: Baseline (Day -1) and Day 2
  Safety and tolerability will be assessed by measuring the clinical laboratory parameters which include hematology, clinical chemistry, routine urinalysis and additional parameters.
Systolic and diastolic blood pressure for each treatment group | Baseline (Day 1 pre-dose) and Day 2 of each treatment period; and Follow-up Visit
  Safety and tolerability will be assessed by measuring vital signs which include systolic and diastolic blood pressure.
Heart rate for each treatment group | Baseline (Day 1 pre-dose) and Day 2 of each treatment period; and Follow-up Visit
  Safety and tolerability will be assessed by measuring vital signs which include heart rate.
12-lead electrocardiogram (ECG) for each treatment group | Baseline (Day 1 pre-dose) and Day 2 of each treatment period; and Follow-up Visit
  Safety and tolerability will be assessed by measuring ECG using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Yang S, Lee L, Mallett S, Ayer J, Wolstenholme A, Pascoe S. A randomized, crossover study to investigate the pharmacokinetics and safety of inhaled fluticasone furoate and umeclidinium, administered separately and in combination via dry powder inhaler in healthy adult volunteers. Adv Ther. 2015 Feb;32(2):157-71. doi: 10.1007/s12325-015-0184-6. Epub 2015 Feb 21. PMID 25700806
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 116524 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116524?search=study&study_ids=116524#rs
- Available data/document: Dataset Specification: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116524 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register